CLINICAL TRIAL: NCT02661048
Title: CyberHeart's Cardiac Arrhythmia Ablation Treatment: Patients With Refractory Ventricular Tachycardia
Brief Title: CyberHeart's Cardiac Arrhythmia Ablation Treatment: Patients With Refractory Ventricular Tachycardia/Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CyberHeart Inc. -001
Record Dates: First submitted 2015-12-22; First posted 2016-01-21 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Tachycardia, Ventricular
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Open label (Experimental): Non-randomized, open label clinical trial that intends to treat 10 subjects with refractory ventricular tachycardia with the CyberHeart system using standard radiosurgical techniques.
  Interventions: Device: CyberHeart System

INTERVENTIONS:
Device: CyberHeart System — The CyberHeart system uses proprietary software to assist the cardiologist to contour ablation targets. Standard radiosurgical techniques are then used to accomplish ablation

SUMMARY:
The objective of this clinical investigation is to evaluate:

1. the safety and efficacy of the CyberHeart System, CardioPlan™ Software and Laptop, in treating patients with refractory ventricular tachycardia (VT) using the CyberKnife® Radiosurgical System.
2. The CyberHeart System performance with respect to the ability to contour myocardial targets that are transferred to the Multi-plan® Treatment Planning Software of the CyberKnife® system for the production and delivery of a safe radiosurgical treatment plan.

Cardiac radiosurgery is a minimally-non invasive, painless, procedure. Tissue ablation can be accomplished precisely.

DETAILED DESCRIPTION:
This study is a prospective, multi-center (2), single arm, open label US-based feasibility study.

The clinical hypothesis for the study is that the CyberHeart treatment approach will be safe and with further study will not be shown to be inferior to current treatment options, may lead to a survival benefit and improved quality of life.

The ablation to be performed with the CyberHeart System will be targeting the anatomical site of the clinically presenting VT. The application site will be determined by morphological criteria on the 12 lead ECG along with anatomical data from MRI or CT scan imaging. Ablation will be performed at the designated location with the intention to produce substrate modification.

The Study will enroll a maximum of 10 patients.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an implantable cardioverter-defibrillator (ICD)
* Patients with ischemic or non-ischemic cardiomyopathy who have had recurrent symptomatic VT that induced ICD shock(s) following catheter ablation and/or antiarrhythmic drug (AAD) therapy.
* 60 years of age or greater.
* Left ventricular ejection fraction ≥ 20%.
* Failure of or ineligible for catheter ablation.

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Patients with idiopathic VT
* Women who are pregnant
* Prior radiation therapy to the thorax
* Active ischemia or other reversible causes of VT
* Active non-cardiovascular illness or systemic infection
* Presence of thrombus in the right atrium or right ventricle on pre-procedure echocardiogram
* Cardiogenic shock
* NYHA (New York Heart Association) Class IV Heart Failure.
* Presence of incessant VT that is hemodynamically unstable.
* Acute heart failure exacerbation.
* Revascularization in the past 90 days.
* Other disease process that is likely to limit survival to less than 12 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Outcome 1 is the Number of participants with Treatment related Serious Adverse Events as assessed by CTCAE v. 4.0 | 12 months (360 days) with Outcome assesment in first 30 days adn in days 31 to 1 year post treatment.
  Outcome 1 is measured by The number of Participants, and the percentage of participants with :
  - Serious Adverse Events; (1) in the first 30 days, (2) in days 31 to 1 year post treatment, both treatment related, and non-treatment related, separately tabulated.

SECONDARY OUTCOMES:
Number of participants with a change in SF-36 Medical Outcomes Health Survey, as compared to pre-treatment questionaire responses | 12 months
  Participants will complete a SF-36 (Short Form-36) Medical Outcomes Survey before treatment and at each post treatment follow-up check. Absolute numeric numbers will be tabulated and percentage change will be calculated
Number of defibrillation shocks as compared to pretreatment occurrence | 12 months
  Defibrillation shocks will be recorded pre-treatment and post treatment at each follow-up visit.
Ventricular arrhythmia episodes, as compared to pretreatment occurrence | 12 months
  The number of ventricular tachycardia episodes that required either anti-tachycardia pacing, or that self-terminated, will be recorded pre- and post treatment.
Left ventricular function post treatment | 12 months
  Left ventricular systolic and diastolic function will be assessed by echocardiography pre- and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claire McCann, Study Director — Varian Medical Systems
Locations (1):
- Texas Cardiac Arrhythmia Research Foundation, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Loo BW Jr, Soltys SG, Wang L, Lo A, Fahimian BP, Iagaru A, Norton L, Shan X, Gardner E, Fogarty T, Maguire P, Al-Ahmad A, Zei P. Stereotactic ablative radiotherapy for the treatment of refractory cardiac ventricular arrhythmia. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):748-50. doi: 10.1161/CIRCEP.115.002765. No abstract available. PMID 26082532